CLINICAL TRIAL: NCT03414684
Title: A Randomized Phase II Trial of Carboplatin With or Without Nivolumab in First-line Metastatic Triple-negative Breast Cancer
Brief Title: Carboplatin +/- Nivolumab in Metastatic Triple Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Sara Tolaney, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-512; CA209-9JX (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2017-12-01; First posted 2018-01-30 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Carboplatin + Nivolumab (Experimental): * Nivolumab is administered every three weeks intravenously
  * Nivolumab dosage is 360mg
  * Carboplatin is administered every three weeks intravenously
  * Carboplatin dosage is pre-determined by the PI
  Interventions: Drug: Carboplatin; Drug: Nivolumab
- Carboplatin (Active Comparator): * Carboplatin is administered every three weeks intravenously
  * Carboplatin dosage is pre-determined by the PI
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Carboplatin — Carboplatin interferes with the development of the genetic material in a cell, which will cause the cancer cells to die.
Drug: Nivolumab — Nivolumab works by attaching to and blocking a molecule called PD-1. PD-1 is a different molecule that can turn off the immune system by interacting with PD-L1 on the cancer cells
  Other Names: Opdivo
  Arms: Carboplatin + Nivolumab

SUMMARY:
This research study is studying a drug called Carboplatin with or without another study drug, Nivolumab as a possible treatment for triple-negative breast cancer that has spread to other parts of the body.

The interventions involved in this study are:

* Carboplatin
* Nivolumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved nivolumab for your specific disease but it has been approved for other uses. The FDA has approved carboplatin as a treatment option for your disease.

The purpose of this research study is to determine how well carboplatin, by itself, or together with nivolumab, works in treating breast cancer that has spread to other parts of the body. Nivolumab is a recently discovered human monoclonal antibody. An antibody is a type of protein that your immune system (the system that defends your body against potentially harmful particles) uses to find and destroy foreign molecules (particles not typically found in your body, such as bacteria and viruses). Scientists can now make antibodies in the laboratory and produce them for the treatment of many different diseases.

Nivolumab works by attaching to and blocking a molecule called PD-1. PD-1 is a different molecule that can turn off the immune system by interacting with PD-L1 on the cancer cell. Nivolumab has been shown in research studies to prevent PD-1 from shutting down the immune system, thus allowing it to recognize and help your body destroy the cancer cells. You are being asked to participate in this study because triple-negative breast cancer has shown elevated rates of PD-L1 expression.

Nivolumab has been used in other research studies and information from those research studies suggests that nivolumab may help shrink or stabilize your triple negative breast cancer in this study

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed invasive breast cancer, with unresectable locally advanced or metastatic disease. Participants without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis from physical examination or radiologic evaluation.
* Estrogen-receptor and progesterone-receptor expression both ≤ 1% by immunohistochemistry (IHC), and HER2-negative status as determined by the current ASCO/CAP guidelines. If a patient has more than one histological result, the most recent sample will be considered for inclusion.
* Participants must have PD-L1 status available at the time of registration. Standard local testing with any PD-L1 antibody that has been validated in a CLIA-certified environment will be acceptable for including patients on trial.. Primary or metastatic samples may be tested for PD-L1 status.
* Participants must have measurable or evaluable disease by RECIST version 1.1.
* Participants must agree to undergo a research biopsy, if tumor is safely accessible, at baseline. Previously collected archival tissue will also be obtained on all participants. For participants for whom newly-obtained samples cannot be provided (e.g. inaccessible or participant safety concern) the archival tissue alone will be acceptable. Tissue needs to be located and availability confirmed at time of registration (See Section 9 for more details). Participants must agree to a mandatory repeat biopsy 3-6 weeks after starting treatment, if tumor is safely accessible. For patients randomized to carboplatin alone who decide to crossover to nivolumab and nab-paclitaxel at time of progression, a mandatory biopsy will be required if tumor is safely accessible prior to initiating crossover treatment; participants must also agree to undergo this biopsy, if applicable.
* Prior chemotherapy: Participants must have received 0 prior chemotherapeutic regimens for metastatic breast cancer. Prior platinum in the neo/adjuvant setting is permissible, if at least 6 months elapsed since the end of adjuvant systemic therapy to the development of metastatic disease. All toxicities related to prior chemotherapy must have resolved to CTCAE v4.0 grade 1 or lower, unless otherwise specified.
* Prior biologic therapy: Prior poly-ADP ribose polymerase (PARP) inhibitors are not allowed in the metastatic setting. Prior PARP inhibitors in the neo/adjuvant setting are permissible, if at least 6 months elapsed since the end of adjuvant systemic therapy to the development of metastatic disease. All toxicities related to prior biologic therapy must have resolved to CTCAE v4.0 grade 1 or lower, unless otherwise specified.
* Prior radiation therapy: Patients may have received prior radiation therapy. Radiation therapy must be completed at least 14 days prior to registration, and all toxicities related to prior radiation therapy must have resolved to CTCAE v4.0 grade 1 or lower, unless otherwise specified in 3.1.10. Patients may not have had >25% of their bone marrow radiated.
* The subject is ≥18 years old.
* ECOG performance status ≤1 (Karnofsky >60%, see Appendix A).
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,500/mcL
  * Platelets ≥100,000/mcL
  * Hemoglobin ≥ 9.0 g/dl
  * Total bilirubin ≤1.5 × institutional upper limit of normal (ULN) (or ≤2.0 x ULN in patients with documented Gilbert's Syndrome)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN or

    ≤5 × institutional ULN for participants with documented liver metastases
  * Serum creatinine ≤1.5 × institutional ULN OR creatinine clearance ≥ 45 mL/min/ 1.73m2 for participants with creatinine levels above institutional ULN.
* Supportive care (e.g. transfusion of red blood cells) is allowed to meet eligibility criteria.
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 2 weeks prior to registration.
* Childbearing potential is defined as: participants who have not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause) and have not undergone surgical sterilization (removal of ovaries and/or uterus).
* Women of childbearing potential (WOCBP) must agree to use an adequate method of contraception. Contraception is required starting with the first dose of study medication through 150 days (5 months) after the last dose of study medication. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established and proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment with nivolumab and 7 months after the last dose of study treatment (i.e., 90 days (duration of sperm turnover) plus the time required for the investigational drug to undergo approximately five half-lives.)
* Participants on bisphosphonates or RANK ligand inhibitors may continue receiving therapy during study treatment.
* The participant must be capable of understanding and complying with the protocol and willing to sign a written informed consent document

Exclusion Criteria:

* Concurrent administration of any other anti-cancer therapy during the course of this study (bisphosphonates and RANK ligand inhibitors are allowed).
* Prior hypersensitivity to platinum chemotherapy or to any of the excipients of platinum or nivolumab therapy.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including pembrolizumab, ipilimumab, and any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms. Participants with a history of treated central nervous system (CNS) metastases are eligible. Treated brain metastases are defined as those without ongoing requirement for corticosteroids, as ascertained by clinical examination and brain imaging (magnetic resonance imaging or CT scan) completed during screening. Any corticosteroid use for brain metastases must have been discontinued without the subsequent appearance of symptoms for ≥7 days prior to registration. Treatment for brain metastases may include whole brain radiotherapy, radiosurgery, surgery or a combination as deemed appropriate by the treating physician. Radiation therapy must be completed at least 7 days prior to registration
* Major surgery within 2 weeks prior to registration. Patients must have recovered from any effects of any major surgery.
* Uncontrolled, significant intercurrent or recent illness including, but not limited to, ongoing or active infection, uncontrolled non-malignant systemic disease, uncontrolled seizures, or psychiatric illness/social situation that would limit compliance with study requirements in the opinion of the treating investigator.
* Participant has a medical condition that requires chronic systemic steroid therapy (> 10 mg of prednisone daily or equivalent) or any other form of immunosuppressive medication (including disease modifying agents) and has required such therapy in the last 2 years. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic therapy.
* Participant has documented history of autoimmune disease or syndrome that currently requires systemic steroids or immunosuppressive agents.
* History or evidence of active, non-infectious pneumonitis or interstitial lung disease.
* Individuals with a history of a second malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years or are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers that have been diagnosed and treated within the past 3 years are eligible: cervical/prostate carcinoma in situ, superficial bladder cancer, non-melanoma cancer of the skin. Patients with other cancers diagnosed within the past 3 years and felt to be at low risk of recurrence should be discussed with the study sponsor to determine eligibility.
* Participant is known to be positive for the human immunodeficiency virus (HIV), HepBsAg, or HCV RNA. HIV-positive participants are ineligible because of the potential for pharmacokinetic interactions of combination antiretroviral therapy with study drugs. In addition, these participants are at increased risk of fatal infections when treated with marrow-suppressive therapy.
* The participant has received a live vaccine within 28 days prior to registration. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine. The use of the inactivated seasonal influenza vaccine is allowed.
* Women who are pregnant or breastfeeding or adults of reproductive potential not employing an adequate method of contraception.
* Childbearing potential is defined as: participants who have not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause) and have not undergone surgical sterilization (removal of ovaries and/or uterus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2026-07-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (10):
- United States (10):
  - The Stamford Hospital, Stamford, Connecticut
  - Eastern Maine Medical Center, Bangor, Maine
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center in clinical affiliation with South Shore Hospital, South Weymouth, Massachusetts
  - Dana-Farber/New Hampshire Oncology-Hematology, Londonderry, New Hampshire
  - Ohio State University, Columbus, Ohio
  - University of Vermont Medical Center, Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on February 12, 2018, and the last patient was enrolled on September 23, 2020.
Pre-assignment Details: 96 patients were assessed for eligibility, and 18 were found to be ineligible. A total of 78 patients were enrolled and randomized.
Groups:
- Arm A: Carboplatin + Nivolumab: * Nivolumab is administered every three weeks intravenously
  * Nivolumab dosage is 360mg
  * Carboplatin is administered every three weeks intravenously
  * Carboplatin dosage is AUC 6
- Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion: * Carboplatin is administered every three weeks intravenously
  * Carboplatin dosage is AUC 6
    * Upon disease progression, patients on Arm B had the opportunity to cross over to receive single-agent nivolumab (pre-amendment), or combination nivolumab plus nab-paclitaxel (post-amendment); patients that were active on the original crossover treatment (nivolumab monotherapy) before the protocol amendment continued to receive nivolumab monotherapy after the amendment, rather than nivolumab plus nab-paclitaxel
Period: First-course Treatment
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Started | 39 (39 patients were randomized to Arm A) | 39 (39 patients were randomized to Arm B)
Started Treatment | 37 | 38
Completed | 0 (There was no completion of treatment, per protocol. Patients were to remain on treatment until: * Disease progression * Complete response (and treated for at least 24 weeks, with at least two treatments occurring beyond the date when the initial CR was declared) * Intercurrent illness * Unacceptable adverse event(s) * Withdrawal of consent * General/specific changes in the patient's condition that render the patient unacceptable for further treatment) | 0 (There was no completion of treatment, per protocol. Patients were to remain on treatment until: * Disease progression * Complete response (and treated for at least 24 weeks, with at least two treatments occurring beyond the date when the initial CR was declared) * Intercurrent illness * Unacceptable adverse event(s) * Withdrawal of consent * General/specific changes in the patient's condition that render the patient unacceptable for further treatment)
Not Completed | 39 | 39
Not completed — Complete response | 0 | 1
Not completed — Intercurrent illness | 1 | 0
Not completed — Progressive Disease | 31 | 32
Not completed — Adverse Event | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — "Patient proceeded with chest wall excision" | 1 | 0
Not completed — "Participant needed palliative radiation, which is not permitted on study" | 0 | 1
Not completed — Still on treatment | 3 | 0
Not completed — Never started protocol therapy | 2 | 1
Period: Crossover Treatment
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Started | 0 | 18
Completed | 0 | 0 (There was no completion of treatment, per protocol. Patients were to remain on treatment until: * Disease progression * Complete response (and treated for at least 24 weeks, with at least two treatments occurring beyond the date when the initial CR was declared) * Intercurrent illness * Unacceptable adverse event(s) * Withdrawal of consent * General/specific changes in the patient's condition that render the patient unacceptable for further treatment)
Not Completed | 0 | 18
Not completed — Progressive disease | 0 | 12
Not completed — Adverse Event | 0 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Still on treatment | 0 | 2

BASELINE CHARACTERISTICS:
Population: 78 patients were enrolled and randomized, but only 75 patients started protocol therapy. The primary analysis population is the treated population, thus baseline characteristics are shown for the 75 patients that started protocol therapy.
Groups:
- Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion: * Carboplatin is administered every three weeks intravenously
  * Carboplatin dosage is AUC 6
    * Upon disease progression, patients on Arm B had the opportunity to cross over to receive single-agent nivolumab (pre-amendment), or combination nivolumab plus nab-paclitaxel (post-amendment); patients that were active on the original crossover treatment (nivolumab monotherapy) continued to receive nivolumab monotherapy rather than nivolumab plus nab-paclitaxel
- Total: Total of all reporting groups
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Continuous [Median (Full Range); unit: years] | 59.1 [27.9 to 75.8] | 59.1 [25.4 to 75.5] | 59.1 [25.4 to 75.8]
Age, Customized [Count of Participants; unit: Participants]
  Age, years: <40 | 1 | 4 | 5
  Age, years: 40-59 | 19 | 16 | 35
  Age, years: >=60 | 17 | 18 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 33 | 36 | 69
  Unknown or Not Reported | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black or African American | 2 | 3 | 5
  Caucasian | 30 | 34 | 64
  More than one race | 1 | 1 | 2
  Other | 3 | 0 | 3
Germline BRCA Status [Count of Participants; unit: Participants]
  gBRCA1 mutation | 1 | 2 | 3
  gBRCA2 mutation | 0 | 1 | 1
  Non-gBRCA1/2 carrier | 36 | 35 | 71
Programmed death-ligand 1 (PD-L1) immunohistochemistry (IHC) Status -- Local [Count of Participants; unit: Participants]
  Positive | 6 | 6 | 12
  Negative | 11 | 12 | 23
  Not done | 20 | 20 | 40
Programmed death-ligand 1 (PD-L1) immunohistochemistry (IHC) Status -- Central, SP142 [Count of Participants; unit: Participants]
  Positive (>=1% IC) | 14 | 14 | 28
  Negative (<1% IC) | 23 | 24 | 47
Stromal tumor-infiltrating lymphocytes (sTILs) [Count of Participants; unit: Participants]
  0% | 1 | 0 | 1
  1-9% | 23 | 19 | 42
  10-49% | 11 | 17 | 28
  >=50% | 1 | 1 | 2
  Unknown | 1 | 1 | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  0-Fully active, able to carry on pre-disease performance without restriction | 28 | 28 | 56
  1-Restricted in strenuous physical activity but able to perform work of a light or sedentary nature | 9 | 10 | 19
Inflammatory breast cancer [Count of Participants; unit: Participants]
  Yes | 1 | 3 | 4
  No | 36 | 35 | 71
Prior anthracycline in neoadjuvant/adjuvant setting [Count of Participants; unit: Participants]
  Yes | 1 | 4 | 5
  No | 36 | 34 | 70
Prior taxane in neoadjuvant/adjuvant setting [Count of Participants; unit: Participants]
  Yes | 9 | 10 | 19
  No | 28 | 28 | 56
Prior platinum in neoadjuvant/adjuvant setting [Count of Participants; unit: Participants]
  Yes | 4 | 3 | 7
  No | 33 | 35 | 68
Number of lines of prior chemotherapy for advanced disease [Count of Participants; unit: Participants]
  0 | 32 | 30 | 62
  1 | 5 | 8 | 13
Baseline lactate dehydrogenase (LDH) [Count of Participants; unit: Participants]
  <= Upper Limit of Normal | 23 | 24 | 47
  > Upper Limit of Normal | 10 | 14 | 24
  Unknown | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Defined as the time from randomization to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation
Time Frame: Assessed from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, up to 3.5 years
Population: The primary efficacy analysis was conducted in the intention-to-treat (ITT) population, which denotes the 62 patients who had 0 prior lines of treatment for advanced disease prior to enrollment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 32 | 30
months | 4.2 [2.7 to 11.5] | 5.5 [4.4 to 19.2]
Statistical Analysis 1: Comparison: Arm A: Carboplatin + Nivolumab vs Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion; Test type: Superiority; p = 0.88, Log Rank; stratified log rank test; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.49 to 1.84] — Reference level is Arm B, such that hazard ratio corresponds to the effect of treatment on Arm A

2. Secondary Outcome: Objective Response Rate by Response Evaluation Criteria in Solid Tumours (RECIST) 1.1
Description: Defined as the percentage of patients achieving a complete response (complete disappearance of all target and non-target lesions; no new lesions) or partial response (at least 30% decrease in the sum of the diameters of target lesions; persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits [i.e., "non-CR/non-PD" in non-target lesions]; and no new lesions) based on RECIST 1.1
Time Frame: Assessed from the start of treatment until disease progression, complete response (after at least 24 weeks of treatment), intercurrent illness, unacceptable toxicity, noncompliance/withdrawal, or general/specific worsening of condition, up to 3.5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 32 | 30
percent of patients | 25.0 [11.5 to 43.4] | 23.3 [9.9 to 42.3]
Statistical Analysis 1: Comparison: Arm A: Carboplatin + Nivolumab vs Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion; Test type: Superiority; p = 1, Fisher Exact; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.29 to 4.18] — Reference level is Arm B, such that the odds ratio corresponds to the effect of treatment on Arm A

3. Secondary Outcome: Objective Response Rate by Immune-Related Response Criteria (irRC)
Description: Defined as the proportion of patients achieving an immune-related complete response (complete disappearance of all target and non-target lesions; no new measurable/unmeasurable lesions) or immune-related partial response (a decrease of the immune-related sum of product diameters [irSPD] of 50% or greater) based on irRC
Time Frame: as for outcome 2
Population: First-course objective response rate by irRC was only evaluated in the 32 patients that received immunotherapy (on Arm A) in the ITT population. Because of this, statistical testing by arm was not performed.
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 32 | 0
percent of patients | 28.1 [13.7 to 46.7] |

4. Secondary Outcome: Overall Survival
Description: Defined as the time from randomization to death due to any cause, or censored at date last known alive
Time Frame: Assessed from date of randomization until the date of death from any cause, up to 3.5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 32 | 30
months | 16.8 [10.4 to NA] — Upper bound inestimable due to insufficient number of events | 11.1 [8.2 to 24.4]
Statistical Analysis 1: Comparison: Arm A: Carboplatin + Nivolumab vs Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion; Test type: Superiority; p = 0.49, Log Rank; stratified log rank test; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.43 to 1.50] — Reference level is Arm B, such that the hazard ratio corresponds to treatment on Arm A

5. Secondary Outcome: Clinical Benefit Rate
Description: Defined as the proportion of patients achieving a complete response or partial response by RECIST 1.1, or stable disease lasting greater than or equal to 24 weeks
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 32 | 30
percent of patients | 34.4 [18.6 to 53.2] | 33.3 [17.3 to 52.8]
Statistical Analysis 1: Comparison: Arm A: Carboplatin + Nivolumab vs Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion; Test type: Superiority; p = 1, Fisher Exact; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.32 to 3.43] — Reference level is Arm B, such that the odds ratio corresponds to treatment on Arm A

6. Secondary Outcome: Duration of Response
Description: Defined as the time measurement criteria are met for CR or PR by RECIST 1.1 (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. Patients without events reported are censored at the last disease evaluation.
Time Frame: Assessed from the time measurement criteria are met for CR or PR by RECIST 1.1 (whichever is first recorded) to the time of first progression, up to 2.75 years
Population: Duration of response was analyzed among the total 15 patients who achieved objective response in the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 8 | 7
months | 19.3 [16.8 to NA] — Upper bound inestimable due to insufficient number of events | 7.7 [2.7 to NA] — Upper bound inestimable due to insufficient number of events
Statistical Analysis 1: Comparison: Arm A: Carboplatin + Nivolumab vs Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion; Test type: Superiority; p = 0.36, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.13 to 2.12] — Reference level is Arm B, such that the hazard ratio corresponds to treatment on Arm A

7. Secondary Outcome: Time to Objective Response
Description: Defined as the time from randomization to the date of the first documented CR or PR by RECIST 1.1, whichever is first recorded
Time Frame: Assessed from randomization to the time of first response, up to 3.5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 32 | 30
months | 4.6 [4.0 to NA] — Upper bound inestimable due to insufficient number of events | 11.2 [4.7 to NA] — Upper bound inestimable due to insufficient number of events
Statistical Analysis 1: Comparison: Arm A: Carboplatin + Nivolumab vs Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion; Test type: Superiority; p = 0.68, Log Rank; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.43 to 3.43] — Reference level is Arm B, such that the hazard ratio corresponds to treatment on Arm A

8. Secondary Outcome: Progression-free Survival Among PD-L1-positive Patients
Description: PFS defined as the time from randomization to the earlier of progression or death due to any cause; participants alive without disease progression are censored at date of last disease evaluation.
  PD-L1 positivity defined as ≥1% of the tumor cell population demonstrating unequivocal staining for PD-L1.
Time Frame: as for outcome 1
Population: A total of 24 patients were PD-L1-positive in the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 13 | 11
months | 8.3 [2.5 to NA] — Upper bound inestimable due to insufficient number of events | 4.7 [1.6 to NA] — Upper bound inestimable due to insufficient number of events
Statistical Analysis 1: Comparison: Arm A: Carboplatin + Nivolumab vs Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion; Test type: Superiority; p = 0.27, Log Rank; stratified log rank test; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.18 to 1.62] — Reference level is Arm B, such that the hazard ratio corresponds to treatment on Arm A

9. Secondary Outcome: Objective Response Rate by RECIST 1.1 Among PD-L1-positive Patients
Description: ORR defined as the proportion of patients achieving a complete response (complete disappearance of all target and non-target lesions; no new lesions) or partial response (at least 30% decrease in the sum of the diameters of target lesions; persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits [i.e., "non-CR/non-PD" in non-target lesions]; and no new lesions) based on RECIST 1.1.
  PD-L1 positivity defined as ≥1% of the tumor cell population demonstrating unequivocal staining for PD-L1.
Time Frame: as for outcome 2
Population: A total of 24 patients were PD-L1-positive in the ITT population.
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 13 | 11
percent of patients | 23.1 [5.0 to 53.8] | 27.3 [6.0 to 61.0]
Statistical Analysis 1: Comparison: Arm A: Carboplatin + Nivolumab vs Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion; Test type: Superiority; p = 1, Fisher Exact; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.08 to 7.78] — Reference level is Arm B, such that the odds ratio corresponds to treatment on Arm A

10. Secondary Outcome: Objective Response Rate by irRC Among PD-L1-positive Patients
Description: ORR by irRC defined as the proportion of patients achieving an immune-related complete response (complete disappearance of all target and non-target lesions; no new measurable/unmeasurable lesions) or immune-related partial response (a decrease of the immune-related sum of product diameters [irSPD] of 50% or greater) based on irRC.
  PD-L1 positivity defined as ≥1% of the tumor cell population demonstrating unequivocal staining for PD-L1.
Time Frame: as for outcome 2
Population: A total of 13 patients were treated with immunotherapy (on Arm A) and were PD-L1-positive in the ITT population. Because first-course irORR was only assessed for patients on Arm A, no statistical testing by arm was performed.
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 13 | 0
percent of patients | 30.8 [9.1 to 61.4] |

11. Secondary Outcome: Overall Survival Among PD-L1-positive Patients
Description: OS defined as the time from randomization to death due to any cause, or censored at date last known alive.
  PD-L1 positivity defined as ≥1% of the tumor cell population demonstrating unequivocal staining for PD-L1.
Time Frame: Assessed from date of randomization until the date of death from any cause, up to 3.5 years
Population: A total of 24 patients were PD-L1-positive in the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 13 | 11
months | 17.6 [4.9 to NA] — Upper bound inestimable due to insufficient number of events | 10.7 [6.7 to NA] — Upper bound inestimable due to insufficient number of events
Statistical Analysis 1: Comparison: Arm A: Carboplatin + Nivolumab vs Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion; Test type: Superiority; p = 0.61, Log Rank; stratified log rank test; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.26 to 2.16] — Reference level is Arm B, such that the hazard ratio corresponds to treatment on Arm A

12. Secondary Outcome: Clinical Benefit Rate Among PD-L1-positive Patients
Description: CBR defined as the proportion of patients achieving a complete response or partial response by RECIST 1.1, or stable disease lasting greater than or equal to 24 weeks.
  PD-L1 positivity defined as ≥1% of the tumor cell population demonstrating unequivocal staining for PD-L1.
Time Frame: as for outcome 2
Population: A total of 24 patients were PD-L1-positive in the ITT population.
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 13 | 11
percent of patients | 30.8 [9.1 to 61.4] | 36.4 [10.9 to 69.2]
Statistical Analysis 1: Comparison: Arm A: Carboplatin + Nivolumab vs Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion; Test type: Superiority; p = 1, Fisher Exact; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.10 to 5.93] — Reference level is Arm B, such that the odds ratio corresponds to treatment on Arm A

13. Secondary Outcome: Duration of Response Among PD-L1-positive Patients
Description: DOR defined as the time measurement criteria are met for CR or PR by RECIST 1.1 (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. Patients without events reported are censored at the last disease evaluation.
  PD-L1 positivity defined as ≥1% of the tumor cell population demonstrating unequivocal staining for PD-L1.
Time Frame: as for outcome 6
Population: Duration of response was assessed only among the 6 PD-L1-positive patients in the ITT population who achieved objective response. Due to insufficient sample size, statistical testing by arm was not performed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 3 | 3
months | 16.8 [NA to NA] — Bounds inestimable due to insufficient sample size/number of events | 4.9 [2.0 to NA] — Upper bound inestimable due to insufficient sample size/number of events

14. Secondary Outcome: Time to Objective Response Among PD-L1-positive Patients
Description: TTOR defined as the time from randomization to the date of the first documented CR or PR by RECIST 1.1, whichever is first recorded.
  PD-L1 positivity defined as ≥1% of the tumor cell population demonstrating unequivocal staining for PD-L1.
Time Frame: Assessed from randomization to the time of first response, up to 3.5 years
Population: A total of 24 patients were PD-L1-positive in the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 13 | 11
months | NA [3.4 to NA] — Median and upper bound inestimable due to insufficient number of responses | NA [3.0 to NA] — Median and upper bound inestimable due to insufficient number of responses
Statistical Analysis 1: Comparison: Arm A: Carboplatin + Nivolumab vs Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion; Test type: Superiority; p = 0.73, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.14 to 3.89] — Reference level is Arm B, such that the hazard ratio corresponds to treatment on Arm A

15. Secondary Outcome: Second-course Progression-free Survival Among Patients Who Crossed Over to Nab-paclitaxel Plus Nivolumab
Description: PFS defined as the time from the start of crossover treatment to the earlier of progression (on crossover therapy) or death due to any cause; participants alive without disease progression are censored at date of last disease evaluation.
Time Frame: Assessed from the start of crossover therapy to the date of first documented progression on crossover therapy or the date of death from any cause, whichever came first, up to 2.8 years
Population: 10 patients in the ITT population who were initially randomized to Arm B (carboplatin monotherapy) crossed over to receive nab-paclitaxel plus nivolumab
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 0 | 10
months |  | 4.1 [1.9 to NA] — Upper bound inestimable due to insufficient sample size / number of events

16. Secondary Outcome: Second-course Objective Response Rate by RECIST 1.1 Among Patients Who Crossed Over to Nab-paclitaxel Plus Nivolumab
Description: ORR defined as the proportion of patients achieving a complete response (complete disappearance of all target and non-target lesions; no new lesions) or partial response (at least 30% decrease in the sum of the diameters of target lesions; persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits [i.e., "non-CR/non-PD" in non-target lesions]; and no new lesions) based on RECIST 1.1., during crossover therapy
Time Frame: Assessed from the start of crossover treatment until disease progression, intercurrent illness, unacceptable toxicity, noncompliance/withdrawal, or general/specific worsening of condition, up to 2.8 years
Population: 10 patients in the ITT population initially randomized to Arm B (carboplatin monotherapy) crossed over to receive nab-paclitaxel plus nivolumab
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 0 | 10
percent of patients |  | 20.0 [2.5 to 55.6]

17. Secondary Outcome: Second-course Objective Response Rate by irRC Among Patients Who Crossed Over to Nab-paclitaxel Plus Nivolumab
Description: ORR by irRC defined as the proportion of patients achieving an immune-related complete response (complete disappearance of all target and non-target lesions; no new measurable/unmeasurable lesions) or immune-related partial response (a decrease of the immune-related sum of product diameters [irSPD] of 50% or greater) based on irRC, during second-course therapy
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 0 | 10
percent of patients |  | 20.0 [2.5 to 55.6]

18. Secondary Outcome: Second-course Clinical Benefit Rate Among Patients Who Crossed Over to Nab-paclitaxel Plus Nivolumab
Description: CBR defined as the proportion of patients achieving a complete response or partial response by RECIST 1.1, or stable disease lasting greater than or equal to 24 weeks, during second course therapy
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 0 | 10
percent of patients |  | 30.0 [6.7 to 65.2]

19. Secondary Outcome: Second-course Duration of Response Among Patients Who Crossed Over to Nab-paclitaxel Plus Nivolumab
Description: DOR defined as the time measurement criteria are met for second-course CR or PR by RECIST 1.1 (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented thereafter. Patients without events reported are censored at the last disease evaluation.
Time Frame: Assessed from the time measurement criteria are met for CR or PR by RECIST 1.1 (whichever is first recorded) on crossover therapy to the time of first progression on crossover therapy, up to 2.5 years
Population: 10 patients in the ITT population initially randomized to Arm B (carboplatin monotherapy) crossed over to receive nab-paclitaxel plus nivolumab, and only 2 of these patients achieved objective response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 0 | 2
months |  | 1.81 [1.81 to NA] — Upper bound inestimable due to insufficient sample size

20. Secondary Outcome: Second-course Time to Objective Response Among Patients Who Crossed Over to Nab-paclitaxel Plus Nivolumab
Description: TTOR defined as the time from start of crossover treatment to the date of the first documented CR or PR by RECIST 1.1 on second-course therapy, whichever is first recorded
Time Frame: Assessed from the start of crossover therapy to the time of first response on crossover therapy, up to 2.8 years
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 0 | 10
months |  | NA [3.5 to NA] — Median and upper bound inestimable due to insufficient number of responses

21. Secondary Outcome: Second-course Overall Survival Among Patients Who Crossed Over to Nab-paclitaxel Plus Nivolumab
Description: Second-course OS defined as the time from the start of crossover treatment to death due from any cause, or censored at date last known alive.
Time Frame: Assessed from the start of crossover therapy until the date of death from any cause, up to 2.8 years
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 0 | 10
months |  | 12.9 [6.4 to NA] — Upper bound inestimable due to insufficient number of events

22. Secondary Outcome: Progression-free Survival Among BRCA-mutant Patients
Description: PFS defined as the time from randomization to the earlier of progression or death due to any cause; participants alive without disease progression are censored at date of last disease evaluation.
  BRCA-mutant patients were those having BRCA1 or BRCA2 mutations.
Time Frame: as for outcome 1
Population: A total of 2 patients in the ITT population had BRCA1 or BRCA2 mutations.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 0 | 2
months |  | 4.74 [4.74 to NA] — Upper bound inestimable due to insufficient sample size/number of events

23. Secondary Outcome: Objective Response Rate by RECIST 1.1 Among BRCA-mutant Patients
Description: ORR defined as the proportion of patients achieving a complete response (complete disappearance of all target and non-target lesions; no new lesions) or partial response (at least 30% decrease in the sum of the diameters of target lesions; persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits [i.e., "non-CR/non-PD" in non-target lesions]; and no new lesions) based on RECIST 1.1.
  BRCA-mutant patients were those with BRCA1 or BRCA2 mutations.
Time Frame: as for outcome 2
Population: A total of 2 patients in the ITT population had BRCA1 or BRCA2 mutations.
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 0 | 2
percent of patients |  | 50.0 [1.3 to 98.7]

24. Secondary Outcome: Objective Response Rate by irRC Among BRCA-mutant Patients
Description: ORR by irRC defined as the proportion of patients achieving an immune-related complete response (complete disappearance of all target and non-target lesions; no new measurable/unmeasurable lesions) or immune-related partial response (a decrease of the immune-related sum of product diameters [irSPD] of 50% or greater) based on irRC.
  BRCA-mutant patients were those with BRCA1 or BRCA2 mutations.
Time Frame: as for outcome 2
Population: There were 0 patients treated with immunotherapy (on Arm A) and had BRCA1 or BRCA2 mutations in the ITT population.
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Overall Survival Among BRCA-mutant Patients
Description: OS defined as the time from randomization to death due to any cause, or censored at date last known alive.
  BRCA-mutant patients were those with BRCA1 or BRCA2 mutations.
Time Frame: From date of randomization until the date of death from any cause, assessed up to 3.5 years
Population: A total of 2 patients in the ITT population had BRCA1 or BRCA2 mutations.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 0 | 2
months |  | 24.4 [NA to NA] — Bounds inestimable due to insufficient sample size/number of events

26. Secondary Outcome: Clinical Benefit Rate Among BRCA-mutant Patients
Description: CBR defined as the percentage of patients achieving a complete response or partial response by RECIST 1.1, or stable disease lasting greater than or equal to 24 weeks.
  BRCA-mutant patients were those with BRCA1 or BRCA2 mutations.
Time Frame: as for outcome 2
Population: A total of 2 patients in the ITT population had BRCA1 or BRCA2 mutations.
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 0 | 2
percent of patients |  | 50.0 [1.3 to 98.7]

27. Secondary Outcome: Duration of Response Among BRCA-mutant Patients
Description: DOR defined as the time measurement criteria are met for CR or PR by RECIST 1.1 (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. Patients without events reported are censored at the last disease evaluation.
  BRCA-mutant patients were those with BRCA1 or BRCA2 mutations.
Time Frame: Assessed from the time measurement criteria are met for CR or PR by RECIST 1.1 (whichever is first recorded) to the time of first progression, up to 3.5 years
Population: Only 1 patient in the ITT cohort that had a BRCA1 or BRCA2 mutation also achieved objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 0 | 1
months |  | 2.04 [NA to NA] — Bounds inestimable due to insufficient sample size/number of events

28. Secondary Outcome: Time to Objective Response Among BRCA-mutant Patients
Description: TTOR defined as the time from randomization to the date of the first documented CR or PR by RECIST 1.1, whichever is first recorded.
  BRCA-mutant patients were those with BRCA1 or BRCA2 mutations.
Time Frame: Assessed from randomization to the time of first response, up to 3.5 years
Population: A total of 2 patients in the ITT population had BRCA1 or BRCA2 mutations.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin, Then Nivolumab +/- Nab-paclitaxel After Progression, Per Physician Discretion
Number analyzed (Participants) | 0 | 2
months |  | 3.2 [3.2 to NA] — Upper bound inestimable due to insufficient sample size/number of events

ADVERSE EVENTS:
Time Frame: Adverse event data were collected on the first day of each cycle of treatment, as well as at the end of treatment, for both arms, up to 3.5 years. Additionally, patients on Arm A and crossover patients (only) had an adverse events assessment 100 days (-15/+30 days) after the last dose of nivolumab, up to 3.5 years.
Description: An SAE is any untoward medical occurrence that:
  * results in death
  * is life-threatening (i.e., participant was at risk of death at the time of the event)
  * requires hospitalization or prolongs existing hospitalization
  * results in persistent/significant disability/incapacity
  * is a congenital anomaly/birth defect
  * is an important medical event (that may not be immediately life-threatening or result in hospitalization but may jeopardize the subject / require intervention)
Groups:
- Arm B: Carboplatin; Arm B: Carboplatin -- Crossover: * Carboplatin is administered every three weeks intravenously
  * Carboplatin dosage is AUC 6
    * Upon disease progression, patients on Arm B had the opportunity to cross over to receive single-agent nivolumab (pre-amendment), or combination nivolumab plus nab-paclitaxel (post-amendment); patients that were active on the original crossover treatment (nivolumab monotherapy) continued to receive nivolumab monotherapy rather than nivolumab plus nab-paclitaxel
Arm/Group | Arm A: Carboplatin + Nivolumab | Arm B: Carboplatin | Arm B: Carboplatin -- Crossover
All-Cause Mortality (participants affected / at risk) | 24/37 | 17/38 | 10/18
Serious Adverse Events (participants affected / at risk) | 10/37 | 11/38 | 6/18
Other Adverse Events (participants affected / at risk) | 37/37 | 38/38 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Carboplatin + Nivolumab (N=37) | Arm B: Carboplatin (N=38) | Arm B: Carboplatin -- Crossover (N=18)
Anemia (Blood and lymphatic system disorders) | 2 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Fever (General disorders) | 1 | 0 | 0
Infusion related reaction (General disorders) | 1 | 0 | 0
Allergic reaction (Immune system disorders) | 1 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 0
Joint infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 1 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 1 | 0
Platelet count decreased (Investigations) | 3 | 1 | 2
White blood cell decreased (Investigations) | 1 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 2 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Flu like symptoms (General disorders) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Carboplatin + Nivolumab (N=37) | Arm B: Carboplatin (N=38) | Arm B: Carboplatin -- Crossover (N=18)
Anemia (Blood and lymphatic system disorders) | 25 | 20 | 8
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3 | 4 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 4 | 0
Hypothyroidism (Endocrine disorders) | 11 | 3 | 2
Blurred vision (Eye disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 3
Colitis (Gastrointestinal disorders) | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 18 | 14 | 4
Diarrhea (Gastrointestinal disorders) | 11 | 7 | 9
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 | 3 | 2
Hemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 5 | 0 | 0
Nausea (Gastrointestinal disorders) | 21 | 26 | 7
Vomiting (Gastrointestinal disorders) | 5 | 8 | 3
Chills (General disorders) | 4 | 0 | 0
Edema limbs (General disorders) | 3 | 5 | 0
Fatigue (General disorders) | 28 | 28 | 11
Fever (General disorders) | 5 | 5 | 5
Infusion related reaction (General disorders) | 8 | 0 | 0
Localized edema (General disorders) | 3 | 0 | 3
Non-cardiac chest pain (General disorders) | 2 | 0 | 0
Pain (General disorders) | 10 | 13 | 4
Infections and infestations - Other, specify (Infections and infestations) | 2 | 0 | 2
Lung infection (Infections and infestations) | 4 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0
Skin infection (Infections and infestations) | 2 | 3 | 0
Upper respiratory infection (Infections and infestations) | 2 | 3 | 0
Urinary tract infection (Infections and infestations) | 4 | 0 | 0
Vaginal infection (Infections and infestations) | 2 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 | 3 | 2
Alkaline phosphatase increased (Investigations) | 6 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 7 | 3 | 3
Blood bilirubin increased (Investigations) | 2 | 0 | 0
Creatinine increased (Investigations) | 2 | 0 | 2
Investigations - Other, specify (Investigations) | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 6 | 5 | 2
Neutrophil count decreased (Investigations) | 20 | 21 | 7
Platelet count decreased (Investigations) | 29 | 20 | 5
Weight loss (Investigations) | 4 | 2 | 2
White blood cell decreased (Investigations) | 10 | 8 | 3
Anorexia (Metabolism and nutrition disorders) | 9 | 6 | 5
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 6 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 0 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 7 | 5 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 12 | 7 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 0 | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 6 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 4 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Dizziness (Nervous system disorders) | 6 | 4 | 0
Headache (Nervous system disorders) | 10 | 10 | 5
Nervous system disorders - Other, specify (Nervous system disorders) | 2 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 15 | 11 | 6
Tremor (Nervous system disorders) | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 11 | 7 | 0
Depression (Psychiatric disorders) | 5 | 3 | 0
Insomnia (Psychiatric disorders) | 10 | 5 | 0
Breast pain (Reproductive system and breast disorders) | 5 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 7 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 | 17 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 0 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 5
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 4 | 2 | 0
Flushing (Vascular disorders) | 2 | 0 | 0
Hot flashes (Vascular disorders) | 5 | 0 | 0
Hypertension (Vascular disorders) | 10 | 6 | 0
Lymphedema (Vascular disorders) | 2 | 2 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 0
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 2 | 0
Cholesterol high (Investigations) | 0 | 2 | 0
INR increased (Investigations) | 0 | 2 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Dysgeusia (Nervous system disorders) | 0 | 3 | 2
Paresthesia (Nervous system disorders) | 0 | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Thromboembolic event (Vascular disorders) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT03414684/Prot_SAP_000.pdf